CLINICAL TRIAL: NCT03742583
Title: Evaluating the Burst Pressure of Simulated Bowel Anastomosis Constructed Using the Reverse Half-Hitch Alternating Post Knots
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Boris Zevin, Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SURG-431-18
Record Dates: First submitted 2018-10-12; First posted 2018-11-15 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Education, Medical; Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Square Knot (Active Comparator)
  Interventions: Other: Square Knot
- Reversing Half-Hitch Alternating Post Knot (Active Comparator)
  Interventions: Other: RHAP Knot

INTERVENTIONS:
Other: Square Knot — Standard square knot
  Arms: Square Knot
Other: RHAP Knot — Reversing half-hitch alternating post knot
  Arms: Reversing Half-Hitch Alternating Post Knot

SUMMARY:
Square knots are the gold standard for hand-tied surgical knots; however, they are difficult to reproduce in deep body cavities and can inadvertently result in slipped knots. The investigators have shown in previous work that the reversing half-hitch alternating post (RHAP) surgical knot is a non-inferior alternative to the square surgical knot based on its tensile strength and performance in limited working spaces. Prior to introducing RHAP knot in routine surgical practice, it is important to objectively demonstrate similar physical characteristics of anastomosis created using RHAP and standard square knots. This study aims to compare the burst pressure of cadaveric porcine small bowel anastomosis constructed using RHAP and standard square knots on a flat surface and in a simulated deep body cavity.

The investigators are conducting a prospective randomized controlled study of novice medical students allocated to proficiency-based training in RHAP and square surgical knots. Knot tying proficiency will be assessed using a knot-tying checklist. Number of repetitions and time required to achieve proficiency will be tracked for each group. Once proficiency has been achieved by participants in RHAP and square knots group, each participant will perform two-hand sewn small bowel anastomosis using cadaveric porcine small bowel. One anastomosis will be performed on a flat surface and the other will be formed in a simulated deep body cavity. Burst pressure of the anastomoses will be tested using a column of water, and results will be compared between groups. Simple descriptive statistics will be performed for both groups. Between group comparisons of knot-tying proficiency and burst pressure will be performed using t-test. Learning curves within each group will be analyzed using paired 1-way ANOVA. SPSS Statistics (v. 21, IBM, New York, USA) will be used for all statistical analysis, with significance set to p<0.05.

The investigators hypothesize that burst pressure of cadaveric porcine small bowel anastomosis will be equivalent for anastomosis constructed using RHAP and standard square knots.

The results of this study will provide further validity evidence in support of RHAP as suitable alternative to the square surgical knots.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate first or second year medical/non-medical student

Exclusion Criteria:

* Third year or greater undergraduate medical student

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Burst pressure (mm Hg) of repaired enterotomies | One session ~2-4 hours
  Once the enterotomy in the porcine small bowel has been repaired by participants with knots according to the randomized intervention arm, blinded evaluators will tie off one end of the bowel and fill the other end with normal saline. Pressure will be applied the bag of normal saline and the pressure at which the repaired enterotomy leaks will be recorded. The pressure will be recorded in mm Hg.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's Unviersity, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No